CLINICAL TRIAL: NCT02038699
Title: A First-in-man Phase I/II Single-agent Open-label Dose-escalation Study of Every Three-week Dosing of Oral ONC201 in Patients With Advanced Cancer and Limited Treatment Options
Brief Title: A First-in-man Phase I/II Study of Oral ONC201 in Patients With Advanced Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Protocol not activated.
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00001
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2014-10

CONDITIONS: Advanced Glioblastoma; Advanced Colorectal Cancer; Advanced Triple-negative Breast Cancer; Advanced Non-small Cell Lung Cancer
MeSH Terms: interventions — TIC10 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ONC201 (Experimental): Oral ONC201 will be administered once every three weeks at various doses.
  Interventions: Drug: ONC201

INTERVENTIONS:
Drug: ONC201 — ONC201 capsules will be administered orally once every three weeks with flat dosing. Dosage will be given according to a modified Fibonacci sequence with the anticipated starting dose being 125 mg.
  Other Names: TIC10

SUMMARY:
ONC201 is a new potential drug that kills cancer cells but not normal cells in laboratory studies. This clinical trial will be the first evaluation of ONC201 in humans and will enroll patients with advanced cancer. This trial includes a phase I portion that will evaluate the safety of ONC201 and the recommended dose for the phase II portion. The phase II portion will evaluate the initial efficacy profile of ONC201 in select types of cancer.

DETAILED DESCRIPTION:
ONC201 (TIC10) is a first-in-class small molecule that inactivates the Ras effector target kinases, Akt and ERK, selectively in tumor, but not normal, cells to safely trigger cancer cell death. The dual inactivation of Akt and ERK by ONC201 results in broad-spectrum cytotoxic activity that includes activation of TRAIL-mediated apoptotic and other downstream antitumor effects to produce a potent antitumor response. The safety margin (ratio of therapeutic dose to lowest dose with a mild adverse event) of ONC201 is at least 10-fold in rats and dogs in GLP toxicology. The efficacy of ONC201 has been consistently demonstrated in multiple in vitro, ex vivo, and in vivo preclinical cancer models. Favorable attributes of ONC201 observed in preclinical models include antitumor efficacy with infrequent administration, broad-spectrum activity independent of mutations or tumor type, orally active, high safety margins, synergistic activity with many approved therapies, highly stable, highly water soluble, and ability to penetrate the blood-brain barrier. In the phase I portion of the trial, the hypothesis is that ONC201 will exhibit an acceptable safety profile in patients with advanced cancer. In the phase II portion of the trial, the hypothesis is that ONC201 will show preliminary signs of efficacy in patients with advanced cancer as defined by endpoints that include progression-free survival, response rate, biomarkers, and overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed glioblastoma multiforme, triple-negative breast cancer, colorectal cancer, or non-small cell lung cancer patients with advanced disease and limited therapeutic options.
2. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, MRI, or calipers by clinical exam. For lymph nodes to be considered measurable, the short axis must be ≥15 mm when assessed by CT scan. All other lesions (or sites of disease), including small lesions (longest diameter <10 mm or pathological lymph nodes with ≥10 to <15 mm short axis), are considered non-measurable disease. Bone lesions, leptomeningeal disease, ascites, pleural/pericardial effusions, lymphangitis cutis/pulmonitis, inflammatory breast disease, and abdominal masses (not followed by CT or MRI), are considered non-measurable. See Section 11 for the evaluation of measurable disease.
3. Patients are eligible for enrollment if they have not had prior chemotherapy, radiotherapy, anticancer therapy, or investigational agent within 28 days prior to the first dose (Week 1, Day 1); 42 days weeks in the case of alkylating agents. Patients are eligible for enrollment if they have had no surgery within 6 weeks prior to the first dose. Any number of prior therapies is allowable.
4. All adverse events Grade > 1 related to prior therapies (chemotherapy, radiotherapy, and/or surgery) must be resolved, except for alopecia.
5. Age ≥18 years.
6. ECOG performance status ≤ 2 (Karnofsky ≥ 60%, see Appendix A).
7. Life expectancy of greater than 10 weeks.
8. Patients must have normal organ and marrow function as defined below:

   * leukocytes ≥ 3,000/mcL
   * absolute neutrophil count ≥ 1,500/mcL
   * platelets ≥ 100,000/mcL
   * hemoglobin > 8.0 mg/dL
   * total bilirubin < 2.0 x upper limit of normal
   * AST (SGOT)/ALT (SGPT) ≤2.5 × upper limit of normal creatinine OR creatinine clearance ≥60 mL/min/1.73 m2 for patients with creatinine levels above normal.
9. The effects of ONC201 on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
10. Tumor specimen (paraffin-embedded block or frozen tissue) from prior resection or biopsy available that is sufficient to perform pharmacodynamic assays (>3 slides for IHC)
11. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who have received bevacizumab therapy.
2. Patients with known brain metastases will be excluded from the phase I portion of the study. In the phase II portion, patients with known CNS metastases will be limited to 20% of the patient population to accrue proportionately. Patients with CNS metastases must be stable after therapy for CNS metastases (such as surgery, radiotherapy or stereotactic radiosurgery) for > 3 month and must be off steroid treatment prior to study enrollment and must have a life expectancy of 3 months or greater to be eligible.
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to ONC201 or its excipients.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements
5. Pregnant women are excluded from this study because ONC201 is novel agent with unknown potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ONC201, breastfeeding should be discontinued if the mother is treated with ONC201.
6. Patients with a known HIV-positive test on combination antiretroviral therapy are ineligible for the initial first-in-man trial because of the potential for pharmacokinetic interactions with ONC201. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
7. Patients with known history of cardiac arrhythmias including atrial fibrillation, tachyarrhythmias or bradycardia will be excluded. Patients receiving therapeutic agents known to prolong QT interval will be excluded. Patients with history of CHF, or MI or stroke in the last 3 months will be excluded. Patients with a history of seizures will be excluded form the initial trial because ONC201 crosses the blood-brain barrier and this may affect their anti-seizure therapy.
8. Active drug use or alcoholism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01 (Estimated); Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
In Phase I, to determine the recommended phase II doses of ONC201. | Participants will be followed for the duration of the study, an expected average of 6 months.
In phase II, Progression-free survival of patients treated with ONC201. | from enrollment until first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Faris, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: Sponsor website. — http://oncoceutics.com